CLINICAL TRIAL: NCT02201589
Title: Proposed Single Center Investigational Device Exemption: Feasibility of Endovascular Repair Of Ascending Aortic Pathologies
Brief Title: Feasibility of Endovascular Repair Of Ascending Aortic Pathologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rodney A. White, MD (Other)
Responsible Party: Sponsor-Investigator, Rodney A. White, MD, Chief, Vascular Surgery, MemorialCare Health System
Organization: MemorialCare Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSIDE:Ascending Thoracic Aorta
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Aortic Dissection; Intramural Hematoma; Penetrating Ulcer; Pseudoaneurysm
Keywords: Lesions in the ascending thoracic aorta
MeSH Terms: conditions — Aortic Dissection; Penetrating Atherosclerotic Ulcer; Aneurysm, False

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Endovascular repair of ascending aorta (Experimental): Endovascular repair with Valiant PS-IDE Stent Graft
  Interventions: Device: Endovascular repair with Valiant PS-IDE Stent Graft

INTERVENTIONS:
Device: Endovascular repair with Valiant PS-IDE Stent Graft — Endovascular stent graft repair of lesions in the ascending thoracic aorta using the Medtronic Valiant PS-IDE (Physician Sponsored-Investigational Device Exemption) Stent Graft System with the Captivia Delivery System

SUMMARY:
The purpose of this study is to investigate the outcome of patients with pathologies of the ascending thoracic aorta (diseases in the great blood vessel or artery that leads away from the heart) including type A aortic dissection, retrograde type A aortic dissection, intramural hematoma, penetrating ulcer or pseudoaneurysm who are suitable for endovascular (within the vessel) repair with the Medtronic Valiant PS-IDE (Physician Sponsored-Investigational Device Exemption) Stent Graft. Type A aortic dissection is a condition where blood passes through the inner lining or between the layers of the blood vessel from a tear in the aortic wall (dissection) in the ascending aorta; a retrograde Type A aortic dissection is a condition where the dissection or tear in the ascending aorta starts from the descending aorta; an intramural hematoma is a collection of clotted blood within the aortic wall; a penetrating ulcer has a plaque or clot within the wall and a pseudoaneurysm is a false aneurysm . If left untreated in any of these conditions, the aorta can enlarge and rupture causing injury or death. The plan for these patients is to repair the ascending thoracic aorta using the Medtronic Valiant PS-IDE Stent Graft with the Captivia Delivery System. The Valiant Captivia has been evaluated worldwide and used extensively in patients with type B (descending) thoracic aortic dissection. Since the dissections in the ascending aortas mirror that of the descending aorta, it is expected that this stent graft will deliver similar performance and endurance in patients with type A aortic dissection. The investigators expect to reroute the blood to the true lumen (the inner space within the blood vessel) by covering the proximal (nearest to the heart) tear with the stent graft. The stent graft is a stent frame made from Nitinol wire and covered with an expandable material made of a polyester material. This new study will determine how well the device works to treat dissections, intramural hematomas, penetrating ulcers and pseudoaneurysms in the ascending thoracic aorta.

DETAILED DESCRIPTION:
This is a prospective study with 20 patients planned to be enrolled. Patients who participate will be followed for 5 years after the surgery in which the stent graft was implanted. This will include the following schedule: A CT with and without contrast and echocardiogram 30 days after the Medtronic device is implanted, CT with and without contrast at 6 and 12 months post procedure and once a year from 2 years thru 5 years after the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a Type A thoracic aortic dissection, retrograde Type A thoracic aortic dissection, intramural hematoma, penetrating ulcer or pseudoaneurysm of the ascending thoracic aorta affecting the area between the Sinus of Valsalva and the innominate artery orifice (with no involvement of the aortic valve) and be considered candidates for endovascular repair;
* Patient must also have at least one cm proximal and distal landing zones in the ascending aorta between 28-44 mm in diameter;
* The patient must be deemed high-risk surgical candidate according to the following established criteria: ASA (American Society of Anesthesiologists) class IV.

Exclusion Criteria:

* Pregnant or pediatric patients (younger than 21 years of age);
* Patients who have a condition that threatens to infect the stent graft/aortic valve prosthesis;
* Patients with allergies to the stent graft material;
* Patients or their legally authorized representatives who do not sign the informed consent;
* Patients with expected survival less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Composite of all cause mortality, re-interventions, surgical conversions, post-procedural strokes and ischemic or hemorrhagic events causing motoric, language or cognitive compromise | Within 30 days of the index procedure
  Mortality, re-interventions, surgical conversions and post-procedure adverse events

SECONDARY OUTCOMES:
A composite of successful delivery and deployment of stent graft, coverage of lesion and/or proximal entry tear, aortic remodeling based on serial imaging, rupture | To 30 days
  Successful deployment covering the entry tear, remodeling of lesion determined by serial CT scans and documentation of ruptures

CONTACTS AND LOCATIONS:
Overall Officials: Rodney A White, M.D., Principal Investigator — LA BioMedical Research Institute at Harbor-UCLA Medical Center; Ali Khoynezhad, M.D. PhD., Principal Investigator — LA BioMedical Research Institute at Harbor-UCLA Medical Center
Locations (3):
- United States (3):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - LAC Harbor-UCLA Medical Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No
share data at scientific meetings and publications